CLINICAL TRIAL: NCT06783517
Title: Evaluation of Hyaluronic Acid in Addition to Xenograft Material in Treatment Peri-implant Bony Defects in Immediate Implant Placement Within Maxillary Esthetic Zone
Brief Title: Evaluation of Hyaluronic Acid in Addition to Xenograft in Immediate Implant Placement Within Maxillary Esthetic Zone
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Rabia Mohamad Dakhil, M.Sc.- Master Degree of Oral Medicine & Clinical Periodontology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0104023OM
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Effect of Putty Form Bone Graft in Immediate Implant Placment
MeSH Terms: interventions — cerabone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate dental implant with cerabone® (Experimental): Comprised of ten patients with hopeless non-restorable maxillary anterior and/or premolar tooth within the esthetic zone will be extracted and replaced by an immediately placed dental implant in conjunction with Bovine bone mineral graft material( cerabone®,Botiss biomaterial) followed by healing abutment.
  Interventions: Procedure: cerabone
- immediate dental implant with cerabone plus® (Active Comparator): Comprised of ten patients with hopeless non-restorable maxillary anterior and/or premolar tooth within the esthetic zone will be extracted and replaced by an immediately placed dental implant in conjunction with Bovine bone mineral with sodium hyaluronate graft material (cerabone®plus,Botiss biomaterial) followed by healing abutment.
  Interventions: Procedure: cerabone®plus

INTERVENTIONS:
Procedure: cerabone — Atraumatic removal of remaining root or tooth will be performed Implant will be placed in fresh socket Bovine bone graft (cerabone®,Botiss biomaterial) will be added to the implant
  Arms: immediate dental implant with cerabone®
Procedure: cerabone®plus — Atraumatic removal of remaining root or tooth will be performed Implant will be placed in fresh socket Bovine bone substitute with sodium hyaluronate graft (cerabone®plus,Botiss biomaterial) will be added to the implant
  Arms: immediate dental implant with cerabone plus®

SUMMARY:
Study design:

The present study will be carried out on twenty patients selected from the department of Oral Medicine, Periodontology, Oral Diagnosis and Radiology, Faculty of Dentistry, Mansoura University for replacement of non restorable maxillary anterior and/or premolar teeth within esthetic zone by immediate implant divided into two groups. A written informed consent will be obtained from all patients before their participation in this study.

Evaluation of study:

All patients will be seen at regular time interval for evaluation at the visit of surgical intervention , follow up of clinical parameter will be recorded monthly then three , six months postoperative and six month after loading(with twelve month follow up study).

1. Clinical evaluation:

   Implant stability evaluation Soft tissue evaluation
2. Radiographic evaluation:

   * Marginal bone loss(MBL).

DETAILED DESCRIPTION:
Study design:

The present study will be carried out on two groups of patients.

A-Patients Sample:

Twenty patients selected from the department of Oral Medicine, Periodontology, Oral Diagnosis and Radiology, Faculty of Dentistry, Mansoura University for replacement of non restorable maxillary anterior and/or premolar teeth within esthetic zone by immediate implant. A written informed consent will be obtained from all patients before their participation in this study.

i. Group (1): Comprised of ten patients with hopeless non-restorable maxillary anterior and/or premolar tooth within the esthetic zone will be extracted and replaced by an immediately placed dental implant in conjunction with Bovine bone mineral graft material( cerabone®,Botiss biomaterial) followed by healing abutment.

ii. Group (2): Comprised of ten patients with hopeless non-restorable maxillary anterior and/or premolar tooth within the esthetic zone will be extracted and replaced by an immediately placed dental implant in conjunction with Bovine bone mineral with sodium hyaluronate graft material (cerabone®plus,Botiss biomaterial) followed by healing abutment.

Inclusion criteria:

• Patients who are medically free from any systemic diseases.

• Patients with good oral hygiene and regular maintenance.

* Age of patients will be >20 years.
* Presence of at least single non restorable maxillary anterior and/or premolar tooth due to caries, root resorption, endodontic failure, root fracture or tooth with open apex.
* No acute infection is present within both periodontal and/or peri-apical area within the tooth of concern and/or adjacent teeth.
* Patients with extraction socket type I.
* Free from history of clenching, tapping and bruxism.
* Patients prepared to co-operate and comply with the follow-up and maintenance program.

Exclusion criteria:

• Patients taking medications known to influence bone metabolism ( such as heparin, warfarin, corticosteroid).

• Smoking and alcoholic patients.

* History of radiation in the head and neck region.
* Insufficient interocclusal distance for implant placement and restoration.
* Patient with lack of stable posterior occlusion.
* Pregnant, lactating and post-menopausal female patients. Complete medical history, dental history will be taken to all of patients in the study.

Materials:

A. Dental Implants: Conventional 2 pieces screw type dental implants. B. Bone substitute: Bovine bone graft material (cerabone®,Botiss biomaterial) and Bovine bone substitute with sodium hyaluronate graft material (cerabone®plus,Botiss biomaterial).

C. Trephine bur: to create intentional bony defect in experimental rabbits. D. Ostell: to measure the primary and secondary stability of the implant.

Methods:

1. Pre-operative measurements:

   A. Photographs: for all items under research. B. Preoperative Radiographs: CBCT will be taken for clinical patients before treatment.

   C. Antibiotic administration for both patients and rabbits before implant placement.
2. Surgical Procedures:

1. Clinical sample (patients) :

• Atraumatic removal of remaining root or tooth will be performed using periotome, appropriate forceps and elevators in an attempt to preserve the buccal plate of bone and soft tissue.

• Implant will be placed in fresh socket using implant motor with saline coolant after curettage and its size is determined according to pre-operative CBCT within both groups.

* Group (1): Bovine bone graft (cerabone®,Botiss biomaterial)will be added to the implant.
* Group (2): Bovine bone substitute with sodium hyaluronate graft (cerabone®plus,Botiss biomaterial) will be added to the implant.
* followed by healing abutment.
* Post-operative care: The patients will be instructed to consume soft food for eight weeks Patients will be maintained on amoxicillin twice a day for six days and Ibuprofen 400mg 2 to 4 times daily
* loading will begin at three to four months from surgical intervention.

  3-Evaluation of study:

A. Patients evaluation:

All patients will be seen at regular time interval for evaluation at the visit of surgical intervention , follow up of clinical parameter will be recorded monthly then three , six months postoperative and six month after loading(with twelve month follow up study).

1. Clinical evaluation:

   i. Soft tissue evaluation: This will be done in both groups where, soft tissue evaluation will be done using probing depth(PD) and pink esthetic score (PES) around dental implant.

   ii. Implant stability evaluation: Using Osstell implant stability will be assessed in both groups soon after implant placement to assess primary implant stability then three , six and twelve months after surgery to assess secondary implant stability.
2. Radiographic evaluation:

   Radiographic assessment will be held preoperative ,six and twelve months after implant placement for evaluation of:

   • Marginal bone loss(MBL).

   Statistical Analysis:

   All data will be collected and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are medically free from any systemic diseases.

  * Patients with good oral hygiene and regular maintenance.
  * Age of patients will be >20 years.
  * Presence of at least single non restorable maxillary anterior and/or premolar tooth due to caries, root resorption, endodontic failure, root fracture or tooth with open apex.
  * No acute infection is present within both periodontal and/or peri-apical area within the tooth of concern and/or adjacent teeth.
  * Patients with extraction socket type I.
  * Free from history of clenching, tapping and bruxism.
  * Patients prepared to co-operate and comply with the follow-up and maintenance program.

Exclusion Criteria:

* • Patients taking medications known to influence bone metabolism ( such as heparin, warfarin, corticosteroid).

  * Smoking and alcoholic patients.
  * History of radiation in the head and neck region.
  * Insufficient interocclusal distance for implant placement and restoration.
  * Patient with lack of stable posterior occlusion.
  * Pregnant, lactating and post-menopausal female patients. Complete medical history, dental history will be taken to all of patients in the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
radiographic marginal bone change | preoperative , at time implant placement, six and twelve months after implant placement
  Radiographic cone beam tomography (CBCT) assessment will be held preoperative ,at time implant placement, six and twelve months after implant placement
Implant stability evaluation | at time of placement, three , six months after surgery to assess secondary implant stability
  Using Osstell implant stability will be assessed in both groups soon after implant placement to assess primary implant stability then three , six months after surgery to assess secondary implant stability

SECONDARY OUTCOMES:
Soft tissue evaluation | monthly then three , six months postoperative and six month after loading
  This will be done in both groups where, soft tissue evaluation will be done using probing depth(PD) and pink esthetic score (PES) around dental implant

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Egypt, Mansora, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peric Kacarevic Z, Kavehei F, Houshmand A, Franke J, Smeets R, Rimashevskiy D, Wenisch S, Schnettler R, Jung O, Barbeck M. Purification processes of xenogeneic bone substitutes and their impact on tissue reactions and regeneration. Int J Artif Organs. 2018 Nov;41(11):789-800. doi: 10.1177/0391398818771530. Epub 2018 Apr 29. PMID 29707988
- [Background] Dos Santos PL, de Molon RS, Queiroz TP, Okamoto R, de Souza Faloni AP, Gulinelli JL, Luvizuto ER, Garcia IR Jr. Evaluation of bone substitutes for treatment of peri-implant bone defects: biomechanical, histological, and immunohistochemical analyses in the rabbit tibia. J Periodontal Implant Sci. 2016 Jun;46(3):176-96. doi: 10.5051/jpis.2016.46.3.176. Epub 2016 Jun 28. PMID 27382506
- [Background] Cohen DJ, Scott KM, Kulkarni AN, Wayne JS, Boyan BD, Schwartz Z. Acellular mineralized allogenic block bone graft does not remodel during the 10 weeks following concurrent implant placement in a rabbit femoral model. Clin Oral Implants Res. 2020 Jan;31(1):37-48. doi: 10.1111/clr.13544. Epub 2019 Oct 10. PMID 31545532
- [Background] Kyyak S, Blatt S, Wiesmann N, Smeets R, Kaemmerer PW. Hyaluronic Acid with Bone Substitutes Enhance Angiogenesis In Vivo. Materials (Basel). 2022 May 27;15(11):3839. doi: 10.3390/ma15113839. PMID 35683136
- [Background] Raines AL, Sunwoo M, Gertzman AA, Thacker K, Guldberg RE, Schwartz Z, Boyan BD. Hyaluronic acid stimulates neovascularization during the regeneration of bone marrow after ablation. J Biomed Mater Res A. 2011 Mar 1;96(3):575-83. doi: 10.1002/jbm.a.33012. Epub 2011 Jan 10. PMID 21254389
- [Background] Zhao N, Wang X, Qin L, Guo Z, Li D. Effect of molecular weight and concentration of hyaluronan on cell proliferation and osteogenic differentiation in vitro. Biochem Biophys Res Commun. 2015 Sep 25;465(3):569-74. doi: 10.1016/j.bbrc.2015.08.061. Epub 2015 Aug 15. PMID 26284973
- [Background] Pilloni A, Bernard GW. The effect of hyaluronan on mouse intramembranous osteogenesis in vitro. Cell Tissue Res. 1998 Nov;294(2):323-33. doi: 10.1007/s004410051182. PMID 9799448
- [Background] Guo J, Guo S, Wang Y, Yu Y. Adipose-derived stem cells and hyaluronic acid based gel compatibility, studied in vitro. Mol Med Rep. 2017 Oct;16(4):4095-4100. doi: 10.3892/mmr.2017.7055. Epub 2017 Jul 21. PMID 28731160
- [Background] Sasaki T, Watanabe C. Stimulation of osteoinduction in bone wound healing by high-molecular hyaluronic acid. Bone. 1995 Jan;16(1):9-15. doi: 10.1016/s8756-3282(94)00001-8. PMID 7742090
- [Background] Pirnazar P, Wolinsky L, Nachnani S, Haake S, Pilloni A, Bernard GW. Bacteriostatic effects of hyaluronic acid. J Periodontol. 1999 Apr;70(4):370-4. doi: 10.1902/jop.1999.70.4.370. PMID 10328647
- [Background] Kawano M, Ariyoshi W, Iwanaga K, Okinaga T, Habu M, Yoshioka I, Tominaga K, Nishihara T. Mechanism involved in enhancement of osteoblast differentiation by hyaluronic acid. Biochem Biophys Res Commun. 2011 Feb 25;405(4):575-80. doi: 10.1016/j.bbrc.2011.01.071. Epub 2011 Jan 23. PMID 21266161
- [Background] Grigolo B, Lisignoli G, Piacentini A, Fiorini M, Gobbi P, Mazzotti G, Duca M, Pavesio A, Facchini A. Evidence for redifferentiation of human chondrocytes grown on a hyaluronan-based biomaterial (HYAff 11): molecular, immunohistochemical and ultrastructural analysis. Biomaterials. 2002 Feb;23(4):1187-95. doi: 10.1016/s0142-9612(01)00236-8. PMID 11791922
- [Background] Knudson CB, Knudson W. Hyaluronan-binding proteins in development, tissue homeostasis, and disease. FASEB J. 1993 Oct;7(13):1233-41. PMID 7691670
- [Background] Bozic D, Catovic I, Badovinac A, Music L, Par M, Sculean A. Treatment of Intrabony Defects with a Combination of Hyaluronic Acid and Deproteinized Porcine Bone Mineral. Materials (Basel). 2021 Nov 11;14(22):6795. doi: 10.3390/ma14226795. PMID 34832196
- [Background] Kammerer PW, Scholz M, Baudisch M, Liese J, Wegner K, Frerich B, Lang H. Guided Bone Regeneration Using Collagen Scaffolds, Growth Factors, and Periodontal Ligament Stem Cells for Treatment of Peri-Implant Bone Defects In Vivo. Stem Cells Int. 2017;2017:3548435. doi: 10.1155/2017/3548435. Epub 2017 Aug 16. PMID 28951742
- [Background] Shi M, Wang C, Wang Y, Tang C, Miron RJ, Zhang Y. Deproteinized bovine bone matrix induces osteoblast differentiation via macrophage polarization. J Biomed Mater Res A. 2018 May;106(5):1236-1246. doi: 10.1002/jbm.a.36321. Epub 2018 Jan 23. PMID 29280261
- [Background] Prohl A, Batinic M, Alkildani S, Hahn M, Radenkovic M, Najman S, Jung O, Barbeck M. In Vivo Analysis of the Biocompatibility and Bone Healing Capacity of a Novel Bone Grafting Material Combined with Hyaluronic Acid. Int J Mol Sci. 2021 May 1;22(9):4818. doi: 10.3390/ijms22094818. PMID 34062885
- [Background] Kyyak S, Pabst A, Heimes D, Kammerer PW. The Influence of Hyaluronic Acid Biofunctionalization of a Bovine Bone Substitute on Osteoblast Activity In Vitro. Materials (Basel). 2021 May 27;14(11):2885. doi: 10.3390/ma14112885. PMID 34072146
- [Background] Yamada M, Egusa H. Current bone substitutes for implant dentistry. J Prosthodont Res. 2018 Apr;62(2):152-161. doi: 10.1016/j.jpor.2017.08.010. Epub 2017 Sep 15. PMID 28927994
- [Background] Covani U, Canullo L, Toti P, Alfonsi F, Barone A. Tissue stability of implants placed in fresh extraction sockets: a 5-year prospective single-cohort study. J Periodontol. 2014 Sep;85(9):e323-32. doi: 10.1902/jop.2014.140175. Epub 2014 May 16. PMID 24835414
- [Background] Chappuis V, Engel O, Shahim K, Reyes M, Katsaros C, Buser D. Soft Tissue Alterations in Esthetic Postextraction Sites: A 3-Dimensional Analysis. J Dent Res. 2015 Sep;94(9 Suppl):187S-93S. doi: 10.1177/0022034515592869. Epub 2015 Jun 30. PMID 26130259
- [Background] Staas TA, Groenendijk E, Bronkhorst E, Verhamme L, Raghoebar GM, Meijer GJ. Does initial buccal crest thickness affect final buccal crest thickness after flapless immediate implant placement and provisionalization: A prospective cone beam computed tomogram cohort study. Clin Implant Dent Relat Res. 2022 Feb;24(1):24-33. doi: 10.1111/cid.13060. Epub 2022 Jan 3. PMID 34981616
- [Background] Chappuis V, Engel O, Reyes M, Shahim K, Nolte LP, Buser D. Ridge alterations post-extraction in the esthetic zone: a 3D analysis with CBCT. J Dent Res. 2013 Dec;92(12 Suppl):195S-201S. doi: 10.1177/0022034513506713. Epub 2013 Oct 24. PMID 24158340
- [Background] Farronato D, Pasini PM, Manfredini M, Scognamiglio C, Orsina AA, Farronato M. Influence of the implant-abutment connection on the ratio between height and thickness of tissues at the buccal zenith: a randomized controlled trial on 188 implants placed in 104 patients. BMC Oral Health. 2020 Feb 17;20(1):53. doi: 10.1186/s12903-020-1037-5. PMID 32066431
- [Background] Noelken R, Moergel M, Pausch T, Kunkel M, Wagner W. Clinical and esthetic outcome with immediate insertion and provisionalization with or without connective tissue grafting in presence of mucogingival recessions: A retrospective analysis with follow-up between 1 and 8 years. Clin Implant Dent Relat Res. 2018 Jun;20(3):285-293. doi: 10.1111/cid.12595. Epub 2018 Mar 24. PMID 29575589
- [Background] Covani U, Ricci M, Bozzolo G, Mangano F, Zini A, Barone A. Analysis of the pattern of the alveolar ridge remodelling following single tooth extraction. Clin Oral Implants Res. 2011 Aug;22(8):820-5. doi: 10.1111/j.1600-0501.2010.02060.x. Epub 2010 Dec 29. PMID 21198897
- [Background] Mazzocco F, Jimenez D, Barallat L, Paniz G, Del Fabbro M, Nart J. Bone volume changes after immediate implant placement with or without flap elevation. Clin Oral Implants Res. 2017 Apr;28(4):495-501. doi: 10.1111/clr.12826. Epub 2016 Mar 14. PMID 26988739
- [Background] Araujo MG, Silva CO, Misawa M, Sukekava F. Alveolar socket healing: what can we learn? Periodontol 2000. 2015 Jun;68(1):122-34. doi: 10.1111/prd.12082. PMID 25867983
- [Background] Elbrashy A, Osman AH, Shawky M, Askar N, Atef M. Immediate implant placement with platelet rich fibrin as space filling material versus deproteinized bovine bone in maxillary premolars: A randomized clinical trial. Clin Implant Dent Relat Res. 2022 Jun;24(3):320-328. doi: 10.1111/cid.13075. Epub 2022 Mar 30. PMID 35353941
- [Background] Huynh-Ba G, Hoders AB, Meister DJ, Prihoda TJ, Mills MP, Mealey BL, Cochran DL. Esthetic, clinical, and radiographic outcomes of two surgical approaches for single implant in the esthetic area: 1-year results of a randomized controlled trial with parallel design. Clin Oral Implants Res. 2019 Aug;30(8):745-759. doi: 10.1111/clr.13458. Epub 2019 Jun 7. PMID 31099929
- [Background] Ebenezer V, Balakrishnan K, Asir RV, Sragunar B. Immediate placement of endosseous implants into the extraction sockets. J Pharm Bioallied Sci. 2015 Apr;7(Suppl 1):S234-7. doi: 10.4103/0975-7406.155926. PMID 26015721
- [Background] Koutouzis T, Adeinat B, Ali A. The influence of abutment macro-design on clinical and radiographic peri-implant tissue changes for guided, placed, and restored implants: A 1-year randomized controlled trial. Clin Oral Implants Res. 2019 Sep;30(9):882-891. doi: 10.1111/clr.13493. Epub 2019 Jun 24. PMID 31180160
- [Background] Fuentealba R, Jofre J. Esthetic failure in implant dentistry. Dent Clin North Am. 2015 Jan;59(1):227-46. doi: 10.1016/j.cden.2014.08.006. Epub 2014 Sep 26. PMID 25434568